CLINICAL TRIAL: NCT01310725
Title: Mid-term Patency of Radial Artery and No Touch Saphenous Vein as Grafts in CABG; A Randomised Controlled Trial.
Brief Title: Evaluation of Graft Material in Coronary Artery Bypass Grafting (CABG)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Örebro County (Other)
Collaborators: Swedish Heart Lung Foundation (Other); Regional Clinical Research (Other)
Responsible Party: University Hospital Orebro, University Hospital Orebro
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: mdr001
Record Dates: First submitted 2011-03-07; First posted 2011-03-08 (Estimated); Last update posted 2011-03-08 (Estimated); Status verified 2010-09

CONDITIONS: Angina Pectoris
Keywords: CABG; LIMA; saphenous vein; radial artery
MeSH Terms: conditions — Angina Pectoris | interventions — Coronary Artery Bypass

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Coronary artery bypass grafting — Bypass of stenoses in coronary arteries using different types os vessels as conduit.

SUMMARY:
The aim of the study is to evaluate the patency in different kinds of vessels used as graft material in coronary artery bypass grafting.

The hypothesis is that vein grafts harvested with a pedicle of surrounding tissue have the same, or better, patency compared to radial grafts and that skeletonisation of the left internal mammary artery does not effect the patency for this graft.

DETAILED DESCRIPTION:
Patients undergoing coronary artery bypass grafting are included in the study.

Each patient receive a radial artery graft and a vein graft harvested with a pedicle of surrounding tissue to the right and left side of the heart respectively. The left internal mammary artery is used for the left anterior descending artery in a skeletonised or non-skeletonised fashion.

The evaluation is made with angiography up to 5 years after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Isolated coronary artery disease embracing all three main branches of the coronary artery tree.

Exclusion Criteria:

* Kidney insufficiency (Creatinine > 120 µmol/L)
* War-farin anticoagulation therapy
* Ejection fraction < 40%
* Repeat operation
* Other concurrent sur-gery
* Signs of reduced circulation in non-dominant hand
* Other severe illness, or if the patient declines to participate.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2004-01; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Functional grafts defined as opened or closed. | Up to 5 years after surgery.

SECONDARY OUTCOMES:
Degree of stenosis in implanted grafts. | Up to 5 years after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Lars Norgren, MD, PhD, Prof., Study Chair — OREBRO UNIVERSITY
Locations (1):
- Dept of Cardiothoracic Surgery, Orebro University Hospital, Örebro, Sweden